CLINICAL TRIAL: NCT04935151
Title: Holmium Laser Enucleation Versus Bipolar Resection in the Management of a Large Volume (> 80 gm) Symptomatic BPH: a Randomised Controlled Trial
Brief Title: HoLEP vs BPRP in the Management of a Large Volume (> 80 gm) Symptomatic BPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSheemy, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC-TBRI-PT563
Record Dates: First submitted 2021-06-06; First posted 2021-06-22 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: BPH With Urinary Obstruction; Male
Keywords: BPH; enucleation; Large Prostate; LUTS; IPSS; quality of life

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- holmium laser enucleation of the prostate (Active Comparator): holmium laser enucleation of the prostate (HoLEP)
  Interventions: Procedure: holmium laser enucleation of the prostate
- bipolar resection of the prostate (Active Comparator): bipolar resection of the prostate (BPEP)
  Interventions: Procedure: Bipolar resection of the prostate

INTERVENTIONS:
Procedure: holmium laser enucleation of the prostate — cystoscopic transurethral enucleation of the prostate using Holmium laser
  Other Names: HoLEP
  Arms: holmium laser enucleation of the prostate
Procedure: Bipolar resection of the prostate — cystoscopic transurethral resection of the prostate using bipolar energy
  Other Names: BPRP
  Arms: bipolar resection of the prostate

SUMMARY:
To compare bipolar resection versus holmium laser enucleation for management of symptomatic large BPH (> 80 gm)

DETAILED DESCRIPTION:
To compare safety and efficacy of bipolar resection (BPRP) versus holmium laser enucleation (HoLEP) for management of symptomatic large BPH (> 80 gm)

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from LUTS secondary to infravesical obstruction from BPH with failed medical treatment
* International Prostate Symptom Score (IPSS) > 13
* a peak urinary flow rate (Qmax) < 15 ml/sec
* a prostate size ≥ 80 gm

Exclusion Criteria:

* presence of a urethral stricture
* neurological disorder
* bladder cancer
* prostate cancer
* previous history of bladder neck surgery or TURP

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-12-04 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
hemoglobin drop postoperatively (gm/dL) | within two hours after surgery
  change in hemoglobin concentration postoperatively vs preoperatively

SECONDARY OUTCOMES:
operative duration in minutes | Time lapsed during surgery
  operative duration
Hospital stay | From time of randomisation up to last day of admission in hospital (in days) up to 30 days
  Hospitalisation starting from day of surgery till the day of discharge from Hospital in days
blood transfusion | during surgery and hospitalisation up to 10 days
  rate of blood transfusion

OTHER OUTCOMES:
complications (percent) | Three years
  All complications
International prostate symptom score (IPSS) | Three years
  an international commonly used score ranging from 0 - 35 (the worst is 35) evaluating voiding and storage urinary symptoms using 7 questions each one is scored from 0 to 5 according to severity of symptom
Quality of life (QoL) | Three years
  section of International prostate symptom score (IPSS) one question scored from 0 up to 6 (6 is worst)
flowmetry | Three years
  rate of flow (ml urine) per second

CONTACTS AND LOCATIONS:
Overall Officials: Mamdouh A Roshdy, M.D, Study Director — Theodor Bilharz research institue
Locations (2):
- Egypt (2):
  - Cairo University Hospitals, Cairo
  - Theodor Bilharz research institute, Giza

IPD SHARING:
Plan to Share IPD: No